CLINICAL TRIAL: NCT00578565
Title: Rituximab for the Treatment of Rheumatoid Arthritis-Associated Interstitial Pneumonia: A Pilot Study
Brief Title: Rituximab in Rheumatoid Arthritis Lung Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eric Matteson (Other)
Collaborators: Genentech, Inc. (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Eric Matteson, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-007133; UL1RR024150 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Rheumatoid Arthritis; Interstitial Pneumonia
Keywords: Rheumatoid Arthritis; Interstitial Pneumonia; Rheumatology; Rituximab
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): open label, all subjects will receive rituximab
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 1000 mg. I.V.on each days 1 and 15 with repeat dosing at 6 months.
  Other Names: Rituxan; MabThera

SUMMARY:
This study will examine the course of patients with progressive rheumatoid arthritis associated interstitial lung disease (RA-ILD) treated with rituximab for safety and progression-free survival at 48 weeks. Safety of rituximab therapy in this disease will be assessed through patient history, physical exams and laboratory parameters.

* Twelve male/or female patient with RA-associated lung disease (6 of each nonspecific interstitial pneumonia (NSIP) and usual interstitial pneumonia (UIP) histological subtype) will be enrolled
* The study involves 12 visits over 48 weeks
* Rituximab will be administered intravenously at Day 1 and Day 15 with repeat dosing at six months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of RA according to the revised 1987 American Rheumatism Association criteria
2. Absence of clinical features suggesting infection, neoplasm, sarcoidosis, interstitial lung disease other than UIP or NSIP, other collagen vascular disease, or exposure to known fibrogenic drugs or environmental factors
3. Diagnosis of progressive interstitial pneumonia of UIP or NSIP subtype, based on the following criteria

   1. Clinical symptoms consistent with interstitial lung disease with onset between 3 months and 36 months prior to screening.
   2. Worsening as demonstrated by any one of the following within the past year:

      * > 10% decrease in Forced Vital Capacity (FVC)
      * increasing infiltrates on chest X-ray or High Resolution Computed Tomography (HRCT), or worsening dyspnea at rest or on exertion
   3. Diagnosis of UIP or NSIP by either of the following:

      * Open or video-assisted thoracic surgery (VATS) lung biopsy showing definite or probable UIP or NSIP
      * HRCT scan showing definite or probable UIP or NSIP AND abnormal pulmonary function tests (reduced FVC or decreased diffusing capacity of carbon monoxide (DLco) or impaired gas exchange at rest or with exercise) AND insidious onset of otherwise unexplained dyspnea or exertion and bibasilar, inspiratory crackles on auscultation
   4. FVC > 50% of predicted value at Screening
   5. DLco >30% of predicted value at Screening

5. No change of disease-modifying anti-rheumatic drug (DMARD) treatment within the last 3 months

Exclusion Criteria:

1. History of clinically significant environmental or drug exposure known to cause pulmonary fibrosis.
2. Forced expiratory volume in one second (FEV1) FEV1/FVC ratio < 0.6 at screening (pre- or post-bronchodilator).
3. Residual volume > 120% predicted at Screening
4. Evidence of active infection
5. Any pulmonary condition other than UIP/NSIP, which, in the opinion of the site principal investigator, is likely to result in the death of the patient within the next year
6. History of unstable or deteriorating cardiac or neurologic disease
7. Pregnancy or lactation
8. Treatment with cyclophosphamide, cyclosporine, interferon gamma or beta, anti-tumor necrosis factor therapy, anti-interleukin 1 (IL1) therapy or with endothelin receptor blockers within the last 8 weeks; experimental therapy for rheumatoid arthritis
9. Creatinine > 1.5 X upper limit of normal range (ULN) at Screening
10. Hematology outside of specified limits: white blood cell (WBC) < 2,500/mm^3 or absolute neutrophil count (ANC) < 1500
11. Hematocrit < 27% or > 59%, platelets < 100,000/mm^3 at screening
12. Positive hepatitis B or C serology
13. Any medical condition, which in the opinion of the site principal investigator, may be adversely affected by the participation in this study
14. History of recurrent significant infection or history of recurrent bacterial infections
15. Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
16. Abnormal neurological examination reflective of central nervous disease, including paresis, cognitive impairment and problems with coordination
17. Current enrollment in another clinical trial
18. Fever (>99.5º F)
19. History of previous rituximab administration
20. Receipt of any vaccine, particularly live viral vaccines, within 4 weeks of first study dose
21. Decreased Immunoglobulin G (IgG) and Immunoglobulin M (IgM) levels (below lower limit of normal range)
22. Present or past malignancy
23. History of severe allergic or anaphylactic reaction to administration of humanized or murine monoclonal antibodies
24. Positive human immunodeficiency virus (HIV) serology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Matteson, M.D., M.P.H., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Mayo Clinic and Brigham and Women's rheumatology outpatient clinics.
Groups:
- Rituximab: open label, all subjects will receive Rituximab 1000 mg. I.V.on each days 1 and 15 with repeat dosing at 6 months
Period: Overall Study
Arm/Group | Rituximab
Started | 10
Completed | 7
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 10
Age Continuous [Mean (Full Range); unit: years] | 64.7 [43 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10
Duration of Rheumatoid Arthritis (RA) [Mean (Full Range); unit: Years] | 13.8 [0.4 to 44]
Duration of Interstitial Lung Disease (ILD) [Mean (Full Range); unit: Years] | 3.2 [0.0 to 7.5]
Histological subtypes of RA-ILD [Number; unit: participants]
  Nonspecific Interstitial Pneumonia (NSIP) | 6
  Usual Interstitial Pneumonia (UIP) | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Diffusion Capacity for Carbon Monoxide (DLco) From Baseline to 48 Weeks
Description: DLco is one pulmonary function measure. For DLco, worsening was defined as decrease of at least 15% and improvement was defined as increase of at least 15%.
Time Frame: baseline, 48 weeks
Population: Three participants of the 10 enrolled withdrew or died before the end of the study.
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 7
participants
  Stable | 4
  Improved | 2
  Worsened | 1

2. Secondary Outcome: Change in Lung Fibrosis Score as Observed on High Resolution Computerized Tomography (HRCT) Scans, From Baseline to 48 Weeks
Description: Three serial HRCT scans of each patient were scored independently and simultaneously by two core radiologists, who were blinded to the sequence in which three scans were obtained (at screening, 24 and 48 weeks). The HRCT scoring sheet scored different domains of abnormality such as, linear opacities, consolidation, ground-glass density, etc. Radiographers reported composite impression based on scoring according to worsening, no worsening or improvement of relevant domains.
Time Frame: baseline, 48 weeks
Population: Three participants of the 10 enrolled withdrew or died before the end of the study.
Measure: Number; unit: participants
Groups:
- Rituximab: open label, all subjects will receive Rituximab 1000 mg. I.V. on each days 1 and 15 with repeat dosing at 6 months
Arm/Group | Rituximab
Number analyzed (Participants) | 7
participants
  Stable | 5
  Improved | 1
  Worsened | 1

3. Secondary Outcome: Assessment of RA Disease Activity Scores as Measured by the DAS28 Score at Baseline and 48 Weeks
Description: The DAS28 score is a measure of RA disease activity calculated using variables such as swollen joint count, the Erythrocyte Sedimentation Rate (ESR) and patient reported assessment of health.
  Using this data, the DAS28 calculation provides a number on a scale from 0-10 indicating the current activity of a patient's RA. A DAS28 score above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity. Remission is achieved by a DAS28 score lower than 2.6.
Time Frame: baseline, 48 weeks
Population: Three participants of the 10 enrolled withdrew or died before the end of the study.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 7
units on a scale
  Baseline | 5.5 [2.2 to 7.3]
  48 Weeks | 3.3 [2.5 to 4.4]

4. Secondary Outcome: Change in RA Disease Activity From Baseline to 48 Weeks Using the DAS28 Score.
Description: as for outcome 3
Time Frame: baseline, 48 weeks
Population: Three participants of the 10 enrolled withdrew or died before the end of the study.
Measure: Mean (Full Range); unit: percentage of change
Arm/Group | Rituximab
Number analyzed (Participants) | 7
percentage of change | -31.8 [-62 to 24]

5. Primary Outcome: Change in Forced Vital Capacity (FVC) From Baseline to 48 Weeks
Description: FVC is one measure of pulmonary function. For FVC, worsening was defined as decrease of at least 10% and improvement was defined as increase of at least 10%.
Time Frame: baseline, 48 weeks
Population: Three participants of the 10 enrolled withdrew or died before the end of the study.
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 7
participants
  Stable | 4
  Improved | 2
  Worsened | 1

6. Secondary Outcome: Percentage of Change in Health Associated Quality of Life From Baseline to 48 Weeks
Description: The percentage change from baseline to week 48 in a participant's perception of the impact of health on his or her quality of life was collected on the Health Assessment Questionnaire (HAQ). The HAQ measures a person's ability to function with arthritis. The questionnaire is divided into 8 categories (Dressing and Grooming, Arising, Eating, Walking, Hygiene, Reach, Grip and Activities) which include several questions for each category. The category score is determined by the highest score of the set of questions for each category. The disability score is determined by adding the scores for all categories and dividing by 8. The disability scale ranges from 0 (best - without any difficulty) to 3 (worst - unable to do much).
Time Frame: baseline, 48 weeks
Population: Three participants of the 10 enrolled withdrew or died before the end of the study.
Measure: Mean (Full Range); unit: percentage of change
Arm/Group | Rituximab
Number analyzed (Participants) | 7
percentage of change | 85.9 [-80 to 300]

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events during the entire study period, approximately 48 weeks.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=10)
Congestive Heart Failure (Cardiac disorders) | 1 (1) — One patient was hospitalized for congestive heart failure at week 5, considered to be unrelated to study drug, and later died at week 32 of complications following a traumatic hip fracture.
Pneumonia and Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient died at week 6 of possible pneumonia and adult respiratory distress syndrome; a causative organism was not recovered.
Traumatic Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) — One patient was hospitalized for congestive heart failure at week 5, considered to be unrelated to study drug, and later died at week 32 of complications following a traumatic hip fracture.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=10)
Infusion reaction (Injury, poisoning and procedural complications) | 1 (1) — One patient had an infusion reaction with the first infusion, and withdrew from the study.

LIMITATIONS AND CAVEATS:
Given the small number of patients, it could not be determined whether patients with nonspecific interstitial pneumonia (NSIP) or usual interstitial pneumonia (UIP) were more likely to respond. Further research is needed in less advanced disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes